CLINICAL TRIAL: NCT02884180
Title: DEXRAR: DEXamethasone in Revision ARthroplasty: A Randomised, Blinded, 2-group Clinical Trial
Brief Title: DEXRAR: DEXamethasone in Revision ARthroplasty
Acronym: DEXRAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study had met its original objectives for the primary endpoint. A transition to a new regulatory system would have introduced additional costs and delays. Therefore, a strategic decision was made to stop before final enrollment.
Sponsor: Daniel Hägi-Pedersen (Other)
Responsible Party: Sponsor-Investigator, Daniel Hägi-Pedersen, Head of research, consultant, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-DHAG-2016; 2016-002769-72 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative
Keywords: Dexamethasone; Arthroplasty, Replacement, Knee; Revision
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Active Comparator): Dexamethasone 24 mg i.v. after start of anaesthesia
  Interventions: Drug: Dexamethasone
- Treatment B (Placebo Comparator): Saline isotonic i.v. after start of anaesthesia
  Interventions: Drug: Saline isotonic

INTERVENTIONS:
Drug: Dexamethasone — A dose of 24 mg dexamethasone given after start of anaesthesia
  Arms: Treatment A
Drug: Saline isotonic — A dose of 6 ml of isotonic saline given after start of anaesthesia
  Arms: Treatment B

SUMMARY:
Trial name: DEXRAR: Dexamethasone in revision arthroplasty: A randomised, blinded, 2-group clinical trial

Trial acronym: DEXRAR

Background: Effective postoperative pain management is essential for the well-being and rehabilitation of the surgical patient. No "gold standard" exists for pain treatment after revision total knee arthroplasty (TKA) and combinations of different medications are used with virtually no evidence for combined analgesic efficacy.

Objectives: The objective is to investigate the analgesic effect and safety of dexamethasone as a single dose after revision-TKA in combination with paracetamol, ibuprofen and local infiltration analgesia

Intervention: The patients are randomised into to groups: A) 24 mg dexamethasone i.v. B) isotonic saline i.v.

Design and trial size: Placebo controlled, parallel 2-group trial with adequate centralised computer-generated allocation sequence and allocation concealment with block size of 12. Blinding of assessor, investigator, caregivers and patients.

Sample size: 108 eligible patients are needed to detect a difference of 11,3 mg morphine for the first 24 h postoperatively with a standard deviation of 20 mg, a type 1 error rate of 0,05 and a type 2 error rate of 0,20.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral, revision-TKA: Total and major partial revisions were included, i.e. revisions including the femoral and/or the tibial component(s).
* Age > 18
* American Society of Anesthesiologists (ASA) physical status classification system ASA 1- 3.
* Body mass index (BMI) > 18 and < 45
* Women in the fertile age (i.e. until one year after menopause) must have negative urine human chorionic gonadotropin (HCG) pregnancy test
* Patients who gave their written informed consent to participating in the trial after having fully understood the contents of the protocol and restrictions.

Exclusion Criteria:

* Patients who cannot cooperate with the trial.
* Concomitant participation in another trial involving medication
* Patients who cannot understand or speak Danish.
* Patients with allergy to medicines used in the trial.
* Patients with daily use of methadone.
* Contraindications against NSAID, for example previous ulcer, heart failure, liver failure, or renal failure (eGRF < 60 ml/kg/1,73m2), known thrombocytopenia (<100 mia/L)
* Patients suffering from alcohol and/or drug abuse - based on the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Morphine consumption the first 24 hours postoperatively | 0-24 hours postoperatively
  Total need for morphine for the first 24 hours postoperatively administered as both patient controlled analgesia (PCA) and supplemental morphine administered at the post-anaesthesia unit the first hour postoperatively

SECONDARY OUTCOMES:
Pain during movement at 6 hours postoperatively (visual analogue scale) | 6 hours postoperatively
  Pain scores (visual analogue scale (VAS)) with active 45 degrees flexion of the knee at 6 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain during movement at 24 hours postoperatively (visual analogue scale) | 24 hours postoperatively
  Pain scores (visual analogue scale (VAS)) with active 45 degrees flexion of the knee at 24 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain at rest at 6 hours postoperatively (visual analogue scale) | 6 hours postoperatively
  Pain scores (visual analogue scale (VAS)) at rest at 6 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain at rest at 24 hours postoperatively (visual analogue scale) | 24 hours postoperatively
  Pain scores (visual analogue scale (VAS)) at rest at 24 hours postoperatively. No pain = 0; worst imaginable pain = 100
Timed up and go test | 24 hours postoperatively
  Time in seconds, for standing up from a chair, walking 3 meters, turning around, walking back to the chair and sit down again
Adverse events | 0 - 24 hours postoperatively
  Number of patients with one or more adverse events in the intervention period (0-24 hours)
Nausea at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of nausea at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Nausea at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of nausea at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Vomiting the first 24 hours postoperatively | 0-24 hours postoperatively
  Number of vomiting episodes (0-24 hours) measured in the periods 0-6 and 6-24 hours postoperatively
Dizziness at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of dizziness at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Dizziness at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of dizziness at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Sedation at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of sedation at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Sedation at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of sedation at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Anti-emetic treatment the first 24 hours postoperatively | 0-24 hours postoperatively
  Consumption of ondansetron in the period 0-24 hours postoperatively

OTHER OUTCOMES:
Quality of sleep (Verbal rating scale) | 24 hours postoperatively
  Level of quality of sleep. Verbal rating scale: very bad, fairly bad, fairly good, very good
Blood sugar level at 6 hours postoperatively | 6 hours postoperatively
  Level of blood sugar af 6 hours postoperatively in mmol/L
Blood sugar level at 24 hours postoperatively | 24 hours postoperatively
  Level of blood sugar at 24 hours postoperatively in mmol/L
Number of patients with need for antibiotic treatment and/or reoperation within 90 days | 0 - 90 days postoperatively
  Number of patients with need for antibiotic treatment and/or reoperation within 90 days after surgery
Serious adverse events | 0-90 days postoperatively
  Serious adverse events (SAE), including death, within 90 days after surgery defined as SAE (according to International Conference on Harmonization (ICH) - good clinical practice (GCP) - guidelines) except "prolongation of hospitalisation"
Days alive and outside hospital within 90 days after surgery | 0-90 days postoperatively
  Days alive and outside hospital within 90 days after surgery
Quality of live, function | Before surgery
  Oxford Knee Score (OKS) before surgery
Quality of live, function | 6 month postoperatively
  Oxford Knee Score (OKS) 6 month after surgery
Quality of live, function | 12 month postoperatively
  Oxford Knee Score (OKS) 12 month after surgery
Quality of live, function | Before surgery
  EuroQol five dimensions 5 point Lipert scale (EQ-5D-5L) before surgery
Quality of live, function | 6 month postoperatively
  EuroQol five dimensions 5 point Lipert scale (EQ-5D-5L) 6 month after surgery
Quality of live, function | 12 month postoperatively
  EuroQol five dimensions 5 point Lipert scale (EQ-5D-5L) 12 month after surgery
Quality of live, function | Before surgery
  Short Form 36 (SF-36) before surgery
Quality of live, function | 6 month postoperatively
  Short Form 36 (SF-36) 6 month after surgery
Quality of live, function | 12 month postoperatively
  Short Form 36 (SF-36) 12 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, MD, Study Chair — Department of Anaesthesiology, Næstved Hospital
Locations (1):
- Næstved Hospital, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No